CLINICAL TRIAL: NCT02932514
Title: Home Use Sensor (HOUSE) Study
Brief Title: Home Use Sensor Study
Acronym: HOUSE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Senseonics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CTP-0025
Record Dates: First submitted 2016-10-05; First posted 2016-10-13 (Estimated); Last update posted 2017-05-22 (Actual); Status verified 2017-05

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Eversense (Senseonics) CGM System (Experimental)
  Interventions: Device: Eversense (Senseonics) Continuous Glucose Monitoring System

INTERVENTIONS:
Device: Eversense (Senseonics) Continuous Glucose Monitoring System — * Evaluate accuracy of Eversense CGM System to SMBG Meter.
  * Compare performance between abdomen and arm insertion sites.
  * Determine the usability of the Eversense System in a home-use setting for 180 days.

SUMMARY:
The purpose of this clinical investigation is to evaluate the accuracy of the Eversense Continuous Glucose Monitoring System (Eversense System) measurements when compared with a Self-monitoring blood glucose (SMBG) meter. The investigation will assess device performance in two insertion locations (abdomen and upper arm), evaluate safety of the Eversense System usage, and assess the usability of the Eversense system in the hands of user at home setting. Changes in HbA1c from baseline will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects, age ≥18 years
2. Clinically confirmed diagnosis of diabetes mellitus for ≥1 year and using insulin by subcutaneous injection or insulin pump.
3. Subject has signed an informed consent form and is willing to comply with protocol requirements

Exclusion Criteria:

1. Female subjects of childbearing capacity (defined as not surgically sterile or not menopausal for ≥ 1 year) who are lactating or pregnant, intending to become pregnant, or not practicing birth control during the course of the study
2. A condition preventing or complicating the placement, operation or removal of the sensor or wearing of transmitter, including upper extremity deformities or skin condition
3. Symptomatic coronary artery disease; unstable angina; myocardial infarction, transient ischemic attack or stroke within 6 months; uncontrolled hypertension (systolic>160 mm HG or diastolic >100 mm Hg at time of screening); current congestive heart failure; history of cardiac arrhythmia (benign PACs and PVCs allowed). Subjects with asymptomatic coronary artery disease (e.g., CABG, stent placement or angioplasty) may participate if negative stress test within 1 year prior to screening and written clearance from cardiologist documented.
4. History of hepatitis B, hepatitis C, or HIV
5. Currently receiving (or likely to need during the study period): immunosuppressant therapy; chemotherapy; anticoagulant/antithrombotic therapy (excluding aspirin); glucocorticoids (excluding ophthalmic or nasal). This exclusion does include the use of inhaled glucocorticoids and the use of topical glucocorticoids (over sensor site only); antibiotics for chronic infection (e.g. osteomyelitis, endocarditis)
6. A condition requiring or likely to require magnetic resonance imaging (MRI)
7. Known topical or local anesthetic allergy
8. Known allergy to glucocorticoids
9. Any condition that in the investigator's opinion would make the subject unable to complete the study or would make it not in the subject's best interest to participate in the study. Conditions include, but are not limited to, psychiatric conditions, known current or recent alcohol abuse or drug abuse by subject history, a condition that may increase the risk of induced hypoglycemia or risk related to repeated blood testing. Investigator will supply rationale for exclusion
10. Participation in another clinical investigation (drug or device) within 2 weeks prior to screening or intent to participate during the study period
11. The presence of any other active implanted device*

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-10; Primary Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Eversense CGM System for Arm and Abdomen Sensors compared to SMBG Meter as determined by Mean Absolute Relative Difference (MARD) calculations. | 180 Days
Usability of the Eversense CGM System over 180 days will be evaluated through Study Questionnaires. | 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Mona Landin-Olsson, M.D., Ph.D, Principal Investigator — Skane University Hospital
Locations (2):
- Sweden (2):
  - Diabetic Center, Sahlgrenska University Hospital, Gothenburg
  - Skåne University Hospital, Lund